CLINICAL TRIAL: NCT00478348
Title: Adequacy of Drainage During Prosthetic Repair of Incisional Abdominal Hernias: a Randomized Controlled Trial.
Brief Title: Should Prosthetic Repair of Incisional Abdominal Hernias be Drain or Not?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, professor of surgery, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DP-2007-CHV-UNIL
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Complications; Hernia
Keywords: Postoperative Complications; Drainage; Infection; Seroma; Hematoma; Recurrence; Abdominal Wall; Hernia; Surgical Mesh
MeSH Terms: conditions — Postoperative Complications; Hernia; Infections; Seroma; Hematoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drain (Other)
  Interventions: Procedure: Prosthetic repair of abdominal incisional hernia
- No drain (Other)
  Interventions: Procedure: Prosthetic repair of abdominal incisional hernia

INTERVENTIONS:
Procedure: Prosthetic repair of abdominal incisional hernia — Rives-Stoppa repair of incisional hernia

SUMMARY:
The purpose of this study is to determine whether drainage after prosthetic repair of incisional abdominal hernias increases or decreases complications such as infection, seromas and hematomas.

DETAILED DESCRIPTION:
Between 3 to 20% of patients who received a midline laparotomy will develop an incisional hernia.

Primary suture of the defect is associated with a recurrence rate between 25 and 50%.Mesh repair is superior with regard to the recurrence (12-20%), but early postoperative complications include infections, hematomas and seromas.

Some advocate the use of drains in order to diminish secretions and complications. Other claim that drains increase the complication's rate.

In the absence of a randomized controlled trial it's not clear whether drainage could influence positively or negatively the occurence of such complications when performing a prosthetic repair of abdominal incisional hernia.

The aim of this study is to answer this question, comparing prospectively two groups of operated patients: the former with drainage and the latter without.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of midline abdominal wall incisional hernia
* Adults of 20 to 80 years old
* ASA I to III
* Inform consent signed by the patient and investigators

Exclusion Criteria:

* Incisional hernia less than 2 cm
* Groin hernia
* Antibiotic treatment before and during hospital admission
* Emergency admission for strangulated incisional hernia
* Immunosuppressing treatment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Evidence of early clinical infection, hematoma, seroma or recurrence confirmed by ultrasonography or/and laboratory findings. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Demartines, MD, Study Chair — Department of Visceral Surgery, University Hospital Center, Lausanne, Switzerland
Locations (1):
- Department of Visceral Surgery, University Hospital Center, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Willemin M, Schaffer C, Kefleyesus A, Dayer A, Demartines N, Schafer M, Allemann P. Drain Versus No Drain in Open Mesh Repair for Incisional Hernia, Results of a Prospective Randomized Controlled Trial. World J Surg. 2023 Feb;47(2):461-468. doi: 10.1007/s00268-022-06725-4. Epub 2022 Dec 15. PMID 36520177